CLINICAL TRIAL: NCT03138239
Title: The Potential Role of Ga-68-PSMA in Staging, Restaging and Monitoring Response in Primary Liver Cancer: Comparison With F-18-FDG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-17-ES-0056-CTIL
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 16 patients diagnosed with HCC (Experimental): * 12 patients will be tested at the stage of diagnosis (staging)
  * 4 patients who have tested at staging, will be tested again after treatment.
  * 4 patients with treatment failure or recurrence.
  Interventions: Radiation: Ga-68-PSMA scan, and PET -CT F-18-FDG

INTERVENTIONS:
Radiation: Ga-68-PSMA scan, and PET -CT F-18-FDG — The patient will do tow mappings on two different days. It should be noted that there is no importance to the order between the two tests on the condition that they be performed within 7-10 days of each other.
  Both tests will be performed with the Discovery 690 camera, which is located at the Nuclear Medicine Institute.
  First test PET-CT with F-18-FDG PET-CT second test with Ga-68-PSMA

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer and the second leading cause of cancer-related deaths in the world. Hepatitis C virus (HCV) is the most common underlying cause of cirrhosis and HCC in the western world.

The staging of the disease is done by combining blood tests and imaging tests. Ultrasound scanning, computed tomograph (CT) and magnetic resonance imaging (MRI) scans are methods based on identifying or significant change in the liver.

Those changes are sometimes difficult to identify, especially when there are changes in liver structure resulting from disease, such as cirrhosis of the liver.

In many cases it is also difficult to detect secondary scattering in anatomical tests, such as identifying a disease in normal size lymph nodes or early skeletal dissociation.

Functional imaging is not based on structural changes, but on the ability to detect changes in the function and properties of the tissue, such as a change in the cell's metabolic consumption or the presence of proteins that characterize the tumor tissue.PET scans can show tumor cell activity (the cancer cells are more aggressive, get more sugar and therefore see more absorption in PET), detect small tumors and metastases outside the liver (because they do a whole body test). To complete this test, a CT scan is also performed on the same device (PET-CT scanner).

There is a new material called prostate-specific mRNA that is marked with gallium isotope (Ga-68-PSMA). It is the substance that is absorbed into the cells of the blood vessels of the tumor. The Ga-68-PSMA is now widely used in the diagnosis of prostate cancer. The new researches also found the possibility of using Ga-68-PSMA in primary liver cancer in patients because of the over-expression of the antigen in the blood vessels.

Therefore, the tests with Ga-68-PSMA and F-18-FDG will complement each other and will give a complete picture of the extent of the disease.

Each patient has individual characteristics of the tumor, and according to the results it will be possible to adapt the test to the patient with the appropriate material for the disease and this will be effective for the decision to treat and follow up.

At the end of the study it will be possible to offer the study participant the appropriate functional imaging test.

ELIGIBILITY:
Inclusion Criteria:

* 16 patients diagnosed with HCC.

Exclusion Criteria:

* Minors under the age of 18
* Pregnant women
* People without primary liver cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-07-02 (Estimated); Primary Completion 2018-07-02 (Estimated); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
Measure the absorption of PET-CT F-18-FDG and of PET -CT Ga-68-PSMA | The duration of the entire study will last about one year.
  Measuring it in patients with primary liver cancer at staging, restaging and monitoring response.

IPD SHARING:
Plan to Share IPD: No